CLINICAL TRIAL: NCT05013307
Title: Baylor Scott and White Sports Concussion Program Clinical Assessment of Sports Exertion Research Proposal
Brief Title: Clinical Assessment of Sports Exertion
Acronym: CASE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Sports Academy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 021-143
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Return to Sport

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CASE (Experimental): In this prospective study the investigators aim to quantify participants' responses to physical activity. Participants will be asked to engage in physical activity, to identify any provocation of symptoms in adolescents ranging from ages 10 to 22 years. Responses to physical activity will be measured through physiologic markers (e.g., blood pressure, heart rate, oxygen saturation, rate of perceived exertion, dyspnea). Additionally, participants will be monitored for any changes in symptoms that occur during or after physical activity as measured by the modified PCSS symptom inventory.
  Interventions: Other: CASE

INTERVENTIONS:
Other: CASE — The Clinical Assessment for Sports Exertion (CASE) addresses the physical performance of athletes by quantifying physiological and symptomatic responses to dynamic exertion. It was developed by clinicians at the Baylor Scott and White Sports Concussion Program in an effort to identify specific system impairments in athletes who were unable to successfully demonstrate readiness for return to play protocols.

SUMMARY:
The Clinical Assessment for Sports Exertion (CASE) addresses the physical performance of athletes by quantifying physiological and symptomatic responses to dynamic exertion. The CASE is highly sport-specific as it tests multiple body positions that mimic requirements typical of individual and contact sports activities including soccer, gymnastics, cheerleading, swimming, and basketball. It was developed by clinicians at the Baylor Scott and White Sports Concussion Program in an effort to identify specific system impairments in athletes who were unable to successfully demonstrate readiness for return to play protocols. Like the other published forms of concussion exertion testing described above, the CASE is a provocative exercise test that may also prove to be useful in making informed return-to-play decisions based upon the athlete's symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* 10-22 years of age who have participated in organized sport activities within the past 12 months
* Diagnosed with a concussion according to international concussion in sport group criteria
* Asymptomatic at rest and must be cleared from return-to-play by a qualified healthcare professional no later than 30 days following clearance

Exclusion Criteria:

* Orthopedic or neurologic, or other limitations
* History of seizures
* Previous or current diagnoses for cardiopulmonary conditions
* Medical diagnosis of diabetes and/or currently on medications for diabetes (e.g., insulin)
* Uncontrolled asthma
* Pregnancy
* Currently experiencing symptoms of COVID-19 or < 7 days since last symptoms
* History of moderate or severe traumatic brain injury defined as a brain injury with an associated Glasgow Coma Scale score of 12 or less
* Symptom score >1 point on initial PCSS intake
* A current diagnosis of and treatment with medication for attention-deficit/hyperactivity disorder, learning disorder, depression, anxiety, or a history of more than 3 prior concussions
* Limited English proficiency
* Currently taking prescription medication for concussion related impairments
* Anticoagulant or antiplatelet use
* History of a medical condition that mimics the signs and symptoms of prolonged concussion symptoms (eg, history of chronic headaches, active migraines, cardiovascular conditions)

Ages: 10 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate (bpm) | through study completion, an average of 1.5 hours
  Using pulse oximeter placed on index finger heart rate will be recorded.
Blood pressure (mmHg) | through study completion, an average of 1.5 hours
  Using a manual cuff and auscultation method diastolic and systolic scores will be recorded.
Oxygen Saturation (%) | through study completion, an average of 1.5 hours
  Using pulse oximeter placed on index finger oxygen saturation will be recorded.
Rate of Perceived Exertion (Borg 6-20) | through study completion, an average of 1.5 hours
  Using Borg Scale, self report measure of exertion will be recorded. A higher number indicates higher exertion.
Self-rated lightheadedness (0-6) | through study completion, an average of 1.5 hours
  On a scale of 0-6, a self report measure of lightheadedness will be recorded. A higher number indicates worse lightheadedness.
Self-rated dyspnea (Modified Borg 0-10) | through study completion, an average of 1.5 hours
  Using Borg scale, self report measure of dyspnea will be recorded. A higher number indicates worse dyspnea.
Heart rate reserve (peak-rest), beats/min-1 | through study completion, an average of 1.5 hours
  Using metabolic cart, heart rate reserve will be recorded via Garmin heart rate strap.

SECONDARY OUTCOMES:
Modified Post-Concussion Symptom Scale (PCSS) (0-6) | through study completion, an average of 1.5 hours
  Using modified PCSS, self report measure of symptoms will be recorded. A high number indicates worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White Sports Therapy and Research, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No